CLINICAL TRIAL: NCT04609592
Title: Pilot Phase 1 Study of Perioperative Peptide Receptor Radionuclide Therapy (PRRT) in Metastatic, WHO Grade 1 or 2, SSTR Positive, Gastroenteropancreatic Neuroendocrine Tumors Who Are Candidates for Cytoreductive Surgery
Brief Title: Study of PRRT in Metastatic, World Health Organization (WHO) Grade 1 or 2, SSTR Positive, GEP-NET Who Are Candidates for Cytoreductive Surgery
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-52341; NET0030 (Other: OnCore); NCI-2021-03448 (Registry Identifier: CTRP)
Record Dates: First submitted 2020-10-23; First posted 2020-10-30 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Gastroenteropancreatic Neuroendocrine Tumor
MeSH Terms: conditions — Gastro-enteropancreatic neuroendocrine tumor | interventions — lutetium Lu 177 dotatate; Disulfides; gallium Ga 68 dotatate; Ga(III)-DOTATOC; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lutathera (Experimental): 2 cycles of 177Lu Dotatate, followed by cytoreductive surgery, followed by additional 177Lu Dotatate (up to 2 cycles) for residual disease as determined by 68Ga DOTA TATE PET/CT
  Interventions: Drug: Lutathera; Drug: Gallium 68 Dotatate; Procedure: Computed Tomography (CT); Procedure: Magnetic Resonance Imaging (MRI); Procedure: PET/CT

INTERVENTIONS:
Drug: Lutathera — 4 administrations of 7.4 gigabecquerel (GBq) (200 mCi) 177Lu Dotatate +/ 10% at the date and time of infusion, accumulative dose of 29.6 GBq (800 mCi). T
  Other Names: lutetium Lu 177 dotatate; (Lu 177)-N-[(4,7,10-Tricarboxymethyl-1,4,7,10- tetraazacyclododec-1-yl) acetyl]-D-phenylalanyl-L-cysteinyl-L-tyrosyl-D-tryptophanyl-L-lysyl-L-threoninyl-Lcysteinyl-L-threonine-cyclic (2-7) disulfide.; 177 Lu-DOTA-octreotate
Drug: Gallium 68 Dotatate — Standard of care, 2 Megabecquerel (MBq)/kg (0.054 mCi/kg) up to 200 MBq (5.4 mCi)
  Other Names: Gallium-68 DOTA-DPhe1, Tyr3-octreotate
Procedure: Computed Tomography (CT) — Medical Imaging
  Other Names: CT Scan
Procedure: Magnetic Resonance Imaging (MRI) — Medical Imaging
Procedure: PET/CT — Medical Imaging
  Other Names: Positron Emission Tomography (PET)

SUMMARY:
The purpose of this study is to learn about the feasibility and safety of using Peptide Receptor Radionuclide Therapy (PRRT) before and after surgical removal of a tumor. PRRT treatment is based on the administration of a radioactive product, 177-Lu DOTA-0-Tyr3-Octreotate (Lutathera®) and its use before and after surgery is thought to increase the overall survival benefit for patients with SSTR-positive gastroenteropancreatic neuroendocrine tumors GEP-NETs.

DETAILED DESCRIPTION:
Primary Objective(s)

* To assess feasibility and safety of combination of perioperative 177Lu Dotatate and cytoreductive surgery in metastatic GEP NETs Secondary Objective(s)
* To assess response rate (RR) after 2 cycles 177Lu Dotatate
* To assess recurrence free survival (RFS) of the overall treatment strategy
* To assess overall survival (OS) of the overall treatment strategy

ELIGIBILITY:
Inclusion Criteria:

1. Metastatic gastroenteropancreatic NET with lymph nodes or liver metastases only.
2. WHO Grade 1 or 2, Ki 67 ≤ 20% (to be confirmed at Stanford)
3. Must be a candidate for cytoreductive surgery with the goal of R1 resection as determined by a multidisciplinary tumor board discussion
4. Measurable disease as determined by RECIST v1.1
5. Confirmed presence of somatostatin receptors on all target lesions as determined by 68Ga DOTA TATE PET scan
6. Patients ≥ 18 years of age.
7. Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 1
8. Appropriate hematologic, liver and kidney function
9. Patients on octreotide long-acting release (LAR) at a fixed dose of 20 mg or 30 mg at 3 to 4 weeks intervals for at least 12 weeks prior to enrollment in the study

Exclusion Criteria:

1. Prior 177Lu Dotatate treatment
2. Any surgery or radiofrequency ablation within 12 weeks prior to enrollment in the study; or prior radioembolization; chemoembolization; or external beam radiation therapy (EBRT) to > 25% of bone marrow, at any time
3. Any chemotherapy or targeted therapy (including everolimus and sunitinib) within 4 weeks prior to enrollment in the study
4. Known brain metastases
5. Known bone or peritoneal metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-03-17 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Measure Complication free Surgery | 6 months
  The feasibility of perioperative 177Lu Dotatate as part of the therapeutic regimen to treat metastatic neuroendocrine tumors (NETs) will be assessed on the basis of number and proportion of participants who undergo 2 cycles of complication free 177Lu Dotatate therapy followed by cytoreductive surgery without complications, expressed as a number without dispersion. Complications are defined as follows.
  * Radiation fibrosis
  * Hepatic fibrosis by histologic diagnosis
  * Hepatic insufficiency
  * Bowel anastamotic leak (if bowel surgery)
  * Distal pancreatic leak (if pancreas surgery)

SECONDARY OUTCOMES:
Response Rate (RR) | 16 weeks
  Response Rate (RR), as defined by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria, will be determined after 2 pre operative cycles of 177Lu Dotatate. RR will be assessed as the sum of complete response (CR) and partial response (PR), and expressed as a number without dispersion. RECIST criteria are:
  * CR = Disappearance of all target lesions
  * PR = ≥ 30% decrease in the sum of the longest diameter of target lesions
  * Response Rate (RR) = CR + PR
  * Progressive disease (PD) = 20% increase in the sum of the longest diameter of target lesions, and/or the appearance of one or more new lesion(s)
  * Stable disease (SD) = Small changes that do not meet any of the above criteria
Recurrence free Survival (RFS) | 1 year
  Recurrence free Survival (RFS) is defined as the number and proportion of participants that remain alive from the start of treatment without relapse or recurrence of disease, expressed as a number without dispersion.
Overall Survival (OS) | 1 year
  Overall survival (OS) is defined as the number and proportion of participants that remain alive from the start of treatment, expressed as a number without dispersion.

CONTACTS AND LOCATIONS:
Overall Officials: Brendan C Visser, MD, Principal Investigator — Stanford Universiy
Locations (1):
- Stanford Cancer Institute Palo Alto, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No